CLINICAL TRIAL: NCT04778657
Title: National Exhaustive Cohort of Hereditary Stomatocytoses and Other Channelopathies Affecting the Red Blood Cell
Acronym: COHSTO
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210274
Record Dates: First submitted 2021-02-26; First posted 2021-03-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-02

CONDITIONS: Stomatocytosis
Keywords: rare genetic disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hereditary stomatocytosis is a heterogeneous group of rare constitutional diseases of dominant transmission in the vast majority of cases. The data concerning their clinical and biological presentation, and their evolution are few, and come from about thirty clinical cases. The constitution of an exhaustive French cohort of hereditary stomatocytosis will improve the establishment of the diagnosis and the management of patients

DETAILED DESCRIPTION:
The patient is prospectively included. The referring hematologist will inform the patient about participation in the cohort, give him the information note and obtain his non-objection agreement to the use of his data for research purposes.

The data will be collected from the medical file of each patient as part of his usual annual follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with a diagnosis of stomatocytosis without age limit
* Patient affiliated or beneficiary of french Social Security
* No objection from the patient or legal representative

Exclusion Criteria:

* Diagnosis of stomatocytosis excluded by ektacytometry and / or genetics
* Patient under guardianship, with curators or legal protection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients for whom the diagnosis of hereditary stomatocytosis has been made or confirmed by ektacytometry
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-05-06 (Actual); Primary Completion 2041-03-01 (Estimated); Study Completion 2041-03-01 (Estimated)

PRIMARY OUTCOMES:
Obtain a description of the clinical and laboratory data of patients at the time of diagnosis of stomatocytosis | Baseline
  Descriptive analysis of clinical and biological data for the diagnosis of stomatocytosis

SECONDARY OUTCOMES:
Determine the proportion of recurrent genetic mutations and private mutations within our cohort | Baseline
  Number of recurrent genetic mutations and private mutations within our cohort
Establish phenotypes-genotypes relationships | through study completion, an average of 15years
  Specify the phenotypic presentation of each mutation and isolate any correlations genotype-phenotype
Describe the appearance of complications | through study completion, an average of 15years
  Rate of occurrence of complications over time
Describe possible new phenotypic presentations of hereditary stomatocytosis | through study completion, an average of 15years
  Description of the phenotypic presentations of hereditary stomatocytosis

CONTACTS AND LOCATIONS:
Overall Officials: Corinne GUITTON, Principal Investigator — APHP
Locations (1):
- AP-HP, Bicêtre Hospital, Pediatrics - Hematology - Reference center for Sickle cell anemia, Thalassemia and other constitutional diseases of the red blood cell, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No